CLINICAL TRIAL: NCT04850066
Title: Evaluation of the Efficacy of an Equine-assisted Intervention on the Psychosocial Adjustment of Adult Patients Hospitalized and Monitored in Psychiatry: a Randomized Controlled Trial.
Brief Title: Equine-assisted Intervention on Psychosocial Adjustment in Patients With Psychiatric Disorders
Acronym: PEGASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Dreux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A00022-53
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Equine-assisted Therapy
Keywords: Psychiatry; Psychosocial adjustment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine-assisted intervention (Experimental): Brief program (3 sessions)
  Interventions: Behavioral: Equine-assisted intervention
- Control (No Intervention): Standard care with treatments as usual

INTERVENTIONS:
Behavioral: Equine-assisted intervention — Usual care including an equine-assisted intervention carried out on foot, next to the horse, in 3 sessions of 3 hours each, spread over 4 weeks. This program is based on self-awareness, communication, assertiveness and adaptability.
  Arms: Equine-assisted intervention

SUMMARY:
The purpose of this study is to assess the efficacy of a brief equine-assisted intervention on the social adjustment, assertiveness, self-esteem and coping strategies in adult patients with psychosocial dysfunction, hospitalized and followed in psychiatry, as compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized in psychiatry with mental disorders lasting for more than 6 months with an EGF score on the Global Evaluation of Psychosocial Functioning scale of between 31 and 60 at the time of inclusion.

Exclusion Criteria:

* acute psychiatric crisis
* severe comorbidities (such as mental retardation, mental deterioration) which could invalidate informed consent or limit patient compliance with the study protocol.
* medical contraindication to equine-assisted therapy (allergy, immunocompromised patients)
* pregnancy
* no affiliation to a social security scheme
* deprivation of liberty by a judicial decision
* wardship
* horse phobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Social adjustment (self reported) | Baseline and 6 months
  Change in the score of the SAS-SR (social adjustment scale -self report) (from 1 (excellent adjustment) to 5 (bad adjustment))
Social adjustment | Baseline and 6 months
  Change in the score of the SAS (social adjustment scale) (from 1 (excellent adjustment) to 5 (bad adjustment))

SECONDARY OUTCOMES:
Assertiveness | Baseline, 2 and 6 months
  Change in the score of the Rathus assertiveness schedule (from -90 (difficulties of assertivity) to +90 (good assertivity))
Self-esteem | Baseline, 2 and 6 months
  Change in the score of the Rosenberg's Self-Esteem scale (from 10 to 40).
Ways of coping | Baseline, 2 and 6 months
  Change in the score of the Ways of coping checklist (from 27 to 108).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Charles PARIS, Principal Investigator — Pôle Santé Mentale - Centre Hospitalier de Dreux; Anne HERON, Study Director — Unité de Recherche Clinique ARC en CIEL - Centre Hospitalier de Dreux
Locations (1):
- Centre Hospitalier Victor Jousselin, Dreux, France